CLINICAL TRIAL: NCT06743113
Title: A Multi-Center, Randomized, Controlled, Cross-Over Study to Evaluate the Effectiveness of Hypoxic Red Blood Cells Processed With the Hemanext ONE® System Versus Conventional Red Blood Cells in Patients With Transfusion Dependent Sickle Cell Anemia
Brief Title: Hypoxic Red Blood Cells in Sickle Cell Anemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hemanext (Industry)
Collaborators: Emory University (Other); University of Connecticut (Other); University of Pittsburgh Medical Center (Other); Johns Hopkins All Children's Hospital (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-CLIN-0017
Record Dates: First submitted 2024-12-12; First posted 2024-12-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Anaemia; Sickle Cell Anemia Crisis; Sickle Cell Anemia in Children; Sickle Cell Anemia (HbSS, or HbSβ-thalassemia0)
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Intervention Model Description: Each enrolled patient will be randomized to treatment with either hypoxic RBCs or conventional RBCs after successful completion of the screening period. After 6 months in the randomized treatment arm, two "Wash Out" transfusions of conventional RBCs will be scheduled. The patient will then "cross-over" into the other treatment arm to complete another 6 months of treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment A (Hypoxic RBCs) (Experimental): Transfusion of hypoxic red blood cells manufactured with Hemanext ONE system
  Interventions: Device: Hemanext ONE System
- Treatment B (Conventional RBCs) (Active Comparator): Transfusion of conventional red blood cells
  Interventions: Device: Conventional RBCs

INTERVENTIONS:
Device: Hemanext ONE System — Hypoxic red blood cells
  Arms: Treatment A (Hypoxic RBCs)
Device: Conventional RBCs — Conventional red blood cells
  Arms: Treatment B (Conventional RBCs)

SUMMARY:
The overall objective of this study is to evaluate the effectiveness and safety of transfusing hypoxic red blood cells manufactured with the Hemanext ONE system in patients with sickle cell anemia. The Hemanext ONE device was cleared through the De Novo process in September 2023.

DETAILED DESCRIPTION:
In this Direct-to-Phase II study, Hemanext Inc. will carry out a prospective, multi-center, single-blind, randomized, cross-over study in patients with Sickle Cell Anemia, comparing the efficacy of transfusion of hypoxic red blood cells (HRBCs) to transfusions with conventional RBCs. The primary efficacy objective is to demonstrate an increase in %HbA between red cell exchange transfusions (RCE) of HRBCs compared to conventional RBCs. The increases in %HbA (normal Hb) from RCE will be accompanied by a concomitant decrease in sickle Hb (%HbS). The persistence of %HbA will allow for a decrease in the volume of RBCs transfused with an overall decrease in the number of units consumed, which in turn can result in an increase in time (number of days) between transfusions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 7 years of age;
2. Are able to provide informed consent, and assent as applicable, to participate in the study;
3. Diagnosis of Sickle Cell Anemia (SCA) (HbSS, HbSβ0 thalassemia) with participation in a chronic transfusion program and have undergone regular transfusions during at least 6 months prior to Screening;
4. Have had an average interval of at least 14 days between RBC transfusions over the past 6 months;
5. If on iron chelation therapy, have been on a stable dose for ≥3 months prior to screening;

Exclusion Criteria:

1. Are not exclusively transfused at the site;
2. Have a diagnosis of HbSC disease, HbSβ+ thalassemia or another SCD variant (excluding HbSS and HbSβ0 thalassemia)
3. Are routinely transfused with washed, packed RBC units;
4. Have received hemoglobin inducers (e.g. erythropoietin) in the 30 days prior to Screening;
5. Are currently being evaluated for gene therapy;
6. Have any clinically significant pulmonary, cardiovascular, endocrine, hepatic, gastrointestinal, renal, infectious, immunological (including significant allo- or auto-immunization) disease, considered not adequately controlled prior to the study;
7. Are a female of child-bearing potential who is pregnant or planning to become pregnant in the next 14 months;
8. Have a history of allo-immunization that cannot be managed by the local blood bank;
9. Patients who, in the opinion of the Investigator, would not be able or willing to comply with the protocol;
10. Is a ward of the state, prisoner, or transient

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
%HbA Rate of Decline | Through study completion, an average of 14 months
  The primary objective is to evaluate the decreased rate of decline of %HbA between post-transfusion RCE and the subsequent pre-transfusion RCE over 6 transfusion cycles in the hypoxic RBC group compared to the conventional group.

SECONDARY OUTCOMES:
Volume of blood transfused | Through study completion, an average of 14 months
  The mean volume of blood per patient transfused with hypoxic RBCs and with standard RBC units will be analyzed and compared
HgbS Rate of Increase | Through study completion, an average of 14 months
  Average rate of increase of the HgbS measurement between automated red cell exchange (RCE) of hypoxic RBCs compared to conventional RBCs.
Incidence rate of vaso-occlusive crisis. | Through study completion, an average of 14 months
  Incidence rate of vaso-occlusive crisis events through the duration of the study
Incidence rate of acute chest syndrome | Through study completion, an average of 14 months
  Incidence rate of acute chest syndrome events accompanied by fever and/or respiratory symptoms through the duration of the study
Duration (days) of any hospitalization for vaso-occlusive crisis | Through study completion, an average of 14 months
  Mean duration (days) of any hospitalization for vaso-occlusive crisis
Intravascular hemolysis | Through study completion, an average of 14 months
  Level of intravascular hemolysis (measured with free plasma hemoglobin) between each procedure, before and after each Red Cell Exchange.
Serum ferritin | Through study completion, an average of 14 months
  Mean change from baseline in serum ferritin
Changes in hepatic iron content | Through study completion, an average of 14 months
  Mean changes in hepatic iron content
Change in QoL | Through study completion, an average of 14 months
  Mean change in QoL, as measured by validated QoL questionnaires
Total hemoglobin before and after RCE | Through study completion, an average of 14 months
  Mean change before and after transfusions of hypoxically stored RBCs compared to that with conventionally stored RBCs.
Total hematocrit before and after RCE | Through study completion, an average of 14 months
  Mean change before and after transfusions of hypoxically stored RBCs compared to that with conventionally stored RBCs.
Red Cell Exchange events | Through study completion, an average of 14 months
  Mean number of RCE events over the course of the study
Safety assessment | Through study completion, an average of 14 months
  Frequency of adverse event reactions and device deficiencies over the course of the study

OTHER OUTCOMES:
Hemoglobin increment from each transfusion | Through study completion, an average of 14 months
  The hemoglobin increment from each transfusion will be determined by calculating the difference between the patient's post-transfusion and pre-transfusion hemoglobin. It will then be corrected for estimated patient blood volume and the amount of Hb transfused

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Novelli, MD, MS, Principal Investigator — University of Pittsburgh Medical Center; Biree Andemariam, MD, Principal Investigator — New England Sickle Cell Institute, University of Connecticut; Laurel Omert, MD, FACS, Principal Investigator — Hemanext Inc.
Locations (6):
- United States (6):
  - New England Sickle Cell Institute, University of Connecticut, Farmington, Connecticut
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No